CLINICAL TRIAL: NCT02930447
Title: Prospective, Randomized, Controlled Study to Evaluate the Benefit of the Use of Autologous Glue Prepared With RegenKit®-Surgery Device in Abdominoplasty
Brief Title: Evaluation of the Benefit of the Use of Autologous Glue Prepared With RegenKit®-Surgery Device in Abdominoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Regen Lab SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-AG-002
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Abdominoplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Autologous glue will be prepared from the patient's own blood with RegenKit®-Surgery device and applied per-operatively by spraying in the undermining region space between fascia and skin.
  Interventions: Device: Autologous glue
- Control group (No Intervention): Patient from the control group will undergo abdominoplasty according to an identical procedure, but without application of autologous glue or any other treatment product before wound closure.

INTERVENTIONS:
Device: Autologous glue — Patients will undergo abdominoplasty according to the procedure routinely used in the Department of Plastic, Reconstructive and Aesthetic Surgery of HUG. At the end of the procedure, patients assigned to the experimental group will be additionally treated with an application of autologous glue prepared with RegenKit®-Surgery in the undermining region space between fascia and skin, just before closure of the surgical wound.
  Arms: Treatment group

SUMMARY:
Autologous glue therapy with platelet-rich plasma (PRP) was reported to improve outcomes in plastic surgery. However, only pilot studies and retrospective uncontrolled trials have reported the potential benefits of autologous glue treatment up to now. Therefore, a larger, blinded, randomized and placebo-controlled clinical trial would be useful to determine whether platelet-rich plasma is safe and effective in abdominoplasty procedures.

Currently, there are pharmacological options such as artificial fibrin glues composed of homologous fibrinogen and animal-derived thrombin. However, these therapeutics present a risk of transmissible diseases and may induce allergic reactions. Therefore, autologous glues, which are fully made of blood components from the patient itself (autologous fibrinogen contained in PRP and autologous thrombin) represents a safe alternative to artificial biological glues.

Regen Lab SA developed RegenKit®-Surgery to prepare autologous PRP, on one hand, and an autologous activated thrombin serum, on the other hand, in a safe and rapid manner. RegenKit®-Surgery is a CE-marked class IIb medical device.

This study, conducted on 56 patients, will evaluate the effects of autologous glue prepared with RegenKit®-Surgery when used in reconstructive abdominoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with an indication for abdominoplasty
* Signature of informed consent form
* Capable of understanding the study's imperatives

Exclusion Criteria:

* Participation -ongoing or in the last two months- in another clinical trial
* Pregnancy or breastfeeding
* Auto-immune disease (e.g. Hashimoto, rheumatoid arthritis, lupus, etc.)
* Hereditary or acquired hematologic disorder (e.g. drepanocytosis, etc.)
* Haemoglobin < 10g/dl
* Haematocrit < 33%
* Hereditary or acquired coagulation disorder (e.g. platelet dysfunction syndrome, critical thrombocytopenia with a platelet count < 150'000/microlitre, impaired coagulation,etc.)
* Systemic disorders such as diabetes, or hepatitis
* Acute infection
* Any active malignancy
* Chemotherapy
* Refusal or incapacity to give Informed Consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time to drain removal | Maximum of 10 days
  Period of time needed until the drain can be removed after surgery

SECONDARY OUTCOMES:
Volume of exsudates coming from the drain daily | Maximum of 10 days
Percentage of patients with post-operative collections after drain removal | 2 weeks after surgery
Reoperation rate | 6 months
Incidence and severity of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Modarressi, MD, Principal Investigator — University Hospital, Geneva

IPD SHARING:
Plan to Share IPD: Undecided